CLINICAL TRIAL: NCT04602104
Title: A Multiple, Randomized, Double-blinded, Controlled Clinical Study of Allogeneic Human Mesenchymal Stem Cell Exosomes (hMSC-Exos) Nebulized Inhalation in the Treatment of Acute Respiratory Distress Syndrome
Brief Title: A Clinical Study of Mesenchymal Stem Cell Exosomes Nebulizer for the Treatment of ARDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai AbelZeta Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEXARDS
Record Dates: First submitted 2020-08-25; First posted 2020-10-26 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-05

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: human mesenchymal stem cell exosomes
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Phase 1: hMSC-Exos low dose (Experimental): hMSC-Exos low-dose group
  Interventions: Biological: low dose hMSC-Exos
- Phase 1: hMSC-Exos medium dose (Experimental): hMSC-Exos medium-dose group
  Interventions: Biological: medium dose hMSC-Exos
- Phase 1: hMSC-Exos high dose (Experimental): hMSC-Exos high-dose group
  Interventions: Biological: high dose hMSC-Exos
- Phase 2: hMSC-Exos dosage 1 (Experimental): basic treatment+hMSC-Exos (a quarter of MTD/day)
  Interventions: Biological: Dosage 1of hMSC-Exos
- Phase 2: hMSC-Exos dosage 2 (Experimental): basic treatment+hMSC-Exos (MTD/day)
  Interventions: Biological: Dosage 2 of hMSC-Exos
- Phase 2: control group (Placebo Comparator): basic treatment+normal saline
  Interventions: Biological: No hMSC-derived exosomes

INTERVENTIONS:
Biological: low dose hMSC-Exos — basic treatment and 7 times aerosol inhalation of hMSC-Exos (2.0*10^8 particles at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7)
  Arms: Phase 1: hMSC-Exos low dose
Biological: medium dose hMSC-Exos — basic treatment and 7 times aerosol inhalation of hMSC-Exos (8.0*10^8 particles at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7)
  Arms: Phase 1: hMSC-Exos medium dose
Biological: high dose hMSC-Exos — basic treatment and 7 times aerosol inhalation of hMSC-Exos (16.0*10^8 particles at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7)
  Arms: Phase 1: hMSC-Exos high dose
Biological: Dosage 1of hMSC-Exos — basic treatment and 7 times aerosol inhalation of hMSC-Exos (a quarter of MTD/day at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7)
  Arms: Phase 2: hMSC-Exos dosage 1
Biological: Dosage 2 of hMSC-Exos — basic treatment and 7 times aerosol inhalation of hMSC-Exos (MTD/day at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7)
  Arms: Phase 2: hMSC-Exos dosage 2
Biological: No hMSC-derived exosomes — basic treatment and 7 times aerosol inhalation of normal saline (at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7)
  Arms: Phase 2: control group

SUMMARY:
To evaluate allogeneic human mesenchymal stem cell exosomes (hMSC-Exos) in the treatment of acute respiratory distress syndrome (ARDS)

DETAILED DESCRIPTION:
According to the 2012 Berlin diagnostic criteria, there are currently more than 3 million ARDS patients worldwide, accounting for about 10% of patients in the intensive care unit (ICU). In recent years, the incidence of ARDS has increased significantly, which has significantly increased the social and economic burden. The impact of ARDS can even be compared with tumors, AIDS or myocardial infarction. There are the basic clinical treatments, such as using various ventilation methods to improve hypoxia and choosing alternative therapies to improve renal insufficiency. Therefore, there is still a lack of specific treatment measures.

Exosomes are naturally occurring nanosized vesicles and comprised of natural lipid bilayers with the abundance of adhesive proteins that readily interact with cellular membranes. Studies have confirmed that MSC-Exos can improve most of the pathological changes caused by lung infection, reduce pulmonary edema, reduce protein exudation, reduce alveolar inflammation, and clear bacterial infections. Thus, it brings new hope for the treatment of ARDS.

The purpose of this study is to evaluate allogeneic human mesenchymal stem cell exosomes (hMSC-Exos) in the treatment of acute respiratory distress syndrome (ARDS)

ELIGIBILITY:
Inclusion Criteria:

1. The subjects themselves or their family members voluntarily participate in this study and sign the informed consent form;
2. 18-70 years old, male or female;
3. Definitely diagnosed as acute respiratory distress syndrome (ARDS) (according to the Berlin definition and diagnostic criteria of ARDS);
4. Course of disease <96 hours after diagnosis;
5. Chest X-ray showed bilateral infiltration with pulmonary edema; no clinical manifestations of left ventricular hypertension, or pulmonary artery wedge pressure (PAOP) ≤18mmHg.

Exclusion Criteria:

1. Patients with severe allergic constitution;
2. Moderate to severe liver failure (children Pugh score > 12);
3. Patients with severe chronic respiratory diseases, PaCO2 > 50mmhg, and need home oxygen therapy;
4. Severe trauma occurred within 14 days before screening;
5. History of malignant tumor (patients with skin basal cell carcinoma in the past can be included);
6. They are undergoing hemodialysis or peritoneal dialysis;
7. The patients who had deep venous thrombosis or pulmonary embolism within 90 days;
8. Acute myocardial infarction occurred within 30 days;
9. Neuromuscular diseases that result in impaired natural ventilation include, but are not limited to, C5 or higher spinal cord injury, amyotrophic lateral sclerosis, Guillain Barre syndrome, and myasthenia gravis;
10. Obesity (BMI > 28);
11. Lung transplantation;
12. Bone marrow transplantation;
13. Active immunosuppression is defined as receiving immunosuppressive drugs or having a medical condition associated with immunodeficiency. These included: 1) HIV (AIDS or CD4 < 200 cells / mm3); 2) chemotherapy within 6 weeks before randomization; 3) immunosuppressive therapy, including maintenance glucocorticoid therapy (> 40) Results: 1) short term systemic steroid therapy (intravenous or oral) for less than 1 week, topical steroid for skin diseases; 4) absolute neutrophil count < 500 / mm3;
14. Patients undergoing extracorporeal circulation support (ECMO) or high frequency oscillatory ventilation;
15. They were not willing to receive lung protective ventilation (minimum tidal volume 6ml / kg pbw) or liquid management treatment;
16. Have a history of epilepsy, need continuous anticonvulsant therapy, or have received anticonvulsant therapy in the past 3 years;
17. The estimated survival time was less than 30 days;
18. Hepatitis B, hepatitis C, AIDS, syphilis patients;
19. Women of childbearing age are pregnant, lactating or pregnant within one year;
20. Those who could not understand the study protocol;
21. According to the judgment of the researchers, there were other situations in which the patients were not suitable to participate in the study (for example, there were factors to reduce the follow-up compliance, and the patients did not receive relevant supportive treatment, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reaction | up to 14 days
  Incidence of adverse reaction
TTCI | up to 28 days
  Time to Clinical improvement
28-day mortality | up to 28 days
  28-day mortality

SECONDARY OUTCOMES:
Murray lung injury score | baseline and Day 1, Day 2, Day 3, Day 4, Day 5, Day6, Day7, Day14, Day28, Day60
  The minimum value is 0 and the maximum are 16. Higher scores mean a worse outcome.
PaO2/FiO2 | baseline and Day 3, Day7, Day14, Day28, Day60
  oxygen index: the ratio of alveolar oxygen partial pressure to fraction of inspired oxygen
SOFA score | baseline and Day 1, Day 2, Day 3, Day 4, Day 5, Day6, Day7, Day14, Day28, Day60
  The minimum value is 0 and the maximum are 48. Higher scores mean a worse outcome.
ApachⅡ score | baseline and Day 1, Day 2, Day 3, Day 4, Day 5, Day6, Day7, Day14, Day28, Day60
  The minimum value is 0 and the maximum are 24. Higher scores mean a worse outcome.
The number of days the survivor was in ICU | up to 60 days
  The number of days the survivor was in ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers